CLINICAL TRIAL: NCT00821223
Title: Comparison of Phacoemulsification Versus Manual Small Incision Cataract Surgery (SICS) : A Randomized Control Trial
Brief Title: Outcome Following Phacoemulsification Versus Small Incision Cataract Surgery (SICS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iladevi Cataract and IOL Research Center (Other)
Responsible Party: Dr. Alpesh Shah, Iladevi Cataract and IOL Research Center, Ahmedabad, India
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 009
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Last update posted 2010-05-19 (Estimated); Status verified 2010-05

CONDITIONS: Visual Outcomes; Quality of Life
Keywords: phacoemulsification; manual small incision cataract surgery; visual acuity; contrast sensitivity; quality of vision
MeSH Terms: interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- manual small incision cataract surgery (Active Comparator): surgical intervention by small incision cataract surgery
  Interventions: Procedure: manual small incision surgery
- phacoemulsification (Other): surgical intervention by phacoemulsification
  Interventions: Procedure: phacoemulsification and SICS; Procedure: phacoemulsification

INTERVENTIONS:
Procedure: phacoemulsification and SICS — SICS with rigid IOL implantation Phaco with foldable IOL implantation
  Other Names: ECCE; Manual SICS
  Arms: phacoemulsification
Procedure: manual small incision surgery
  Other Names: exrtracapsular cataract surgery
  Arms: manual small incision cataract surgery
Procedure: phacoemulsification — cataract surgery
  Other Names: extracapsualr cataract surgery
  Arms: phacoemulsification

SUMMARY:
Hypothesis :

Phacoemulsification is superior to SICS with regards to:

* Immediate unaided high and low contrast visual performance
* Its impact on quality of life.

DETAILED DESCRIPTION:
Phacoemulsification procedure

* Infiniti Vision System with Software 2.03 or higher, OZil handpiece (HP)
* Anaesthesia: topical
* Incision: temporal clear corneal 2.2 mm single plane
* CCC and hydrodissection, sculpting and division using step by step chop in situ and lateral separation, I/A.
* Single-piece AcrySof IOL (SN60WF) in the bag

SICS procedure

* Anaesthesia: peribulbar
* Incision: superior scleral tunnel 6.5 to 7 mm
* CCC and hydrodissection
* Nuclear expression: blumenthal technique using anterior chamber maintainer, manual cortical clean-up
* Single-piece PMMA (MZ60BD) in the bag

ELIGIBILITY:
Inclusion Criteria:

* Prospective subjects should be diagnosed with senile cataract. Subject must require extraction of cataract in one eye followed by implantation of an AcrySof (SN60WF) or PMMA (MZ60BD) posterior chamber intraocular lens.
* Pupil dilation equal or greater to 7 mm after mydriasis.
* Patients undergoing cataract surgery for the first eye.
* Visual prognosis equal or greater to 6/12.

Exclusion Criteria:

* Patients with history of ocular pathology, glaucoma, uveitis, high myopia, PEX, or corneal pathology.
* Patients with traumatic, subluxated and posterior polar cataract.
* Patients who had previously ocular surgery in the past 6 months prior to the screening visit.
* Patients with diabetic retinopathy.
* Patients who are not suitable for follow-up visits.
* Patients with Fuchs' Dystrophy, Macular Degeneration, Ocular Surface Disease that will interfere with normal recovery.
* Any patients with significant intra-operative complications will be removed from the overall analysis of the results. All patient data should still be recorded, even if from the "excluded" patient group.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2009-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
immediate unaided and aided visual acuity | immediate and mid term (12 months)

SECONDARY OUTCOMES:
Assessment of unaided and aided low contrast sensitivity | 3 and 12 months
Intra-operative complications immediate post-operative day corneal edema anterior chamber inflammation | day 1, 1 week
To assess improvement in quality of life | 3 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alpesh R Shah, Dr, Principal Investigator — Iladevi Cataract and IOL Research Center
Locations (1):
- S. K. Red Cross Eye Hospital,, Dholka, Gujarat, India

REFERENCES:
- [Result] Gogate P, Deshpande M, Nirmalan PK. Why do phacoemulsification? Manual small-incision cataract surgery is almost as effective, but less expensive. Ophthalmology. 2007 May;114(5):965-8. doi: 10.1016/j.ophtha.2006.08.057. Epub 2007 Feb 12. PMID 17296230
- [Result] Ruit S, Tabin G, Chang D, Bajracharya L, Kline DC, Richheimer W, Shrestha M, Paudyal G. A prospective randomized clinical trial of phacoemulsification vs manual sutureless small-incision extracapsular cataract surgery in Nepal. Am J Ophthalmol. 2007 Jan;143(1):32-38. doi: 10.1016/j.ajo.2006.07.023. Epub 2006 Sep 5. PMID 17188040